CLINICAL TRIAL: NCT05989399
Title: Evaluation of Circulating Neutrophils in Antisynthetase Syndrome: a Multicenter Retrospective Study
Brief Title: Evaluation of Circulating Neutrophils in Antisynthetase Syndrome
Acronym: NEUTROSAS2
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI083
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Antisynthetase Syndrome
MeSH Terms: conditions — Antisynthetase syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASyS patients: Patients with antisynthetase syndrome
  Interventions: Diagnostic Test: circulating neutrophils

INTERVENTIONS:
Diagnostic Test: circulating neutrophils — evaluation of circulating neutrophils level

SUMMARY:
Antisynthetase syndrome (ASyS) is a rare and heteregeneous overlapping connective tissue disease, characterized by myositis, interstitial lung disease (ILD), joint involvement, Raynaud's phenomenon and cutaneous manifestations ("mechanic's hands"). Over 50% of patients develop ILD, which is the leading cause of death.

The role of neutrophils - innate immune cells involved in inflammatory processes and induced in particular by cytokines of the Th17 pathway - during AS is unknown. Direct pathogenic role of neutrophils has been described during idiopathic inflammatory myopathies, with an increase of netosis correlated with disease activity and muscle damage. During ASyS, a higher number of alveolar neutrophils has been observed in patients with rapidly progressive ILD.

There are few data on the specific evaluation of circulating neutrophils in ASyS. Investigators suppose that circulating neutrophils level could represent a simple and accessible severity biomarker in patients with ASyS.

The main objective is to evaluate the diagnostic performance of the circulating neutrophils level (> 7000/mm3) at diagnosis on ASyS severity.

The secondary objectives are:

* to define a threshold for circulating neutrophils levels at diagnosis allowing to predict ASyS severity and to assess the diagnostic performance of this threshold.
* to study the correlation between the level of circulating neutrophils and ASyS severity at diagnosis of the disease.
* to compare the circulating neutrophils level at ASyS diagnosis and after 1 year of treatment.
* to compare patients characteristics according to ASyS severity at diagnosis.
* to compare BAL fluid neutrophils level according to ILD severity at ASyS diagnosis in patients with ILD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASyS diagnosis according to Connors criteria

Exclusion Criteria:

* Active infection at ASyS diagnosis
* Evolutive cancer at ASyS diagnosis
* Corticosteroid therapy initiation before circulating neutrophils evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ASyS diagnosis between January 2010 and December 2022
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
circulating neutrophils level > 7000/mm3 | baseline (J0)
number of patients with global severity | baseline (J0)
  global severity defined as presence of severe ILD (PaO2 < 600 mmHg or rapidly progressive ILD), and/or presence of severe myositis (bedrest, or MMT8 score < 30, or MRC muscle testing < 3/5, or swallowing disorers, or dysphagia) and/or presence of myocarditis on cardiac MRI

SECONDARY OUTCOMES:
circulating neutrophils level | baseline (J0)
FVC | baseline (J0)
  FVC percentage
DLCO | baseline (J0)
  DLCO percentage
grade of MRC muscle testing | baseline (J0)
CK level | baseline (J0)
circulating neutrophils level | 12 months
BAL fluid neutrophils level | baseline (J0)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Decker, MD, Principal Investigator — CHU NANCY
Locations (1):
- CHU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No